CLINICAL TRIAL: NCT04783714
Title: Investigating the Effects of a Novel Nutraceutical Combination (Swisse Nutra+ Cholesterol Balance) on Low-density Lipoprotein Cholesterol and Other Markers of Cardiometabolic Health in Australian Adults With Hypercholesterolaemia: A Randomised, Double-blind, Placebo Controlled Trial
Brief Title: Investigating Effects of a Novel Nutraceutical on Hypercholesterolaemia in Australian Adults
Acronym: CLoNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swisse Wellness Pty Ltd (Industry)
Collaborators: Commonwealth Scientific & Industrial Research Organisation (Other); BIONAP SRL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNC-001
Record Dates: First submitted 2021-02-11; First posted 2021-03-05 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-04

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; low-density lipoprotein; nutraceutical; bergamot; artichoke; phytosterols; hydroxytyrosol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Treatment arm and Placebo arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Experimental): Active treatment comprises of 3 soft gel capsules daily (with food) of Swisse Nutra+ Cholesterol Balance, a novel combination nutraceutical containing bergamot juice extract, artichoke leaf extract, hydroxytyrosol and plant sterols, totaling a daily dose of 375 mg bergamot juice extract, 150 mg artichoke leaf extract, 50 mg hydroxytyrosol and 1.8 g sunflower phytosterols.
  Each capsule contains 125mg of bergamot juice extract, 50mg artichoke leaf extract, 16.67mg hydroxytyrosol and 600mg plant sterols.
  The intervention will be administered for 4 months (112 days).
  Interventions: Dietary Supplement: Swisse Nutra+ Cholesterol Balance
- Placebo (Placebo Comparator): 3 soft gel capsules of matching placebo daily (total daily dose of 696 mg palm olein and 232 mg olive oil).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Swisse Nutra+ Cholesterol Balance — Swisse Nutra+ Cholesterol Balance is a multi-ingredient nutraceutical composition contained in a brown soft-gel capsule format. Three capsules are required per dose.Swisse Nutra+ Cholesterol Balance is a multi-ingredient formulation containing artichoke extract, bergamot juice extract, hydroxytyrosol, an antioxidant derived from olive oil and sunflower oil-derived phytosterols. All ingredients target cholesterol reduction by different and complementing mechanisms, as evidenced by human clinical trials. These ingredients have been chosen to work synergistically to alleviate hypercholesterolemia and/or dyslipidemia through multiple pathways, whereby each ingredient works via a different mechanism to lower LDL-cholesterol in the body.
  Arms: Active Group
Dietary Supplement: Placebo — Matched brown soft-gel capsule placebo containing olive oil and palm olein - no therapeutic benefit.
  Arms: Placebo

SUMMARY:
To evaluate the effects of daily consumption of 3 capsules of Swisse Nutra+ Cholesterol Balance on serum LDL-cholesterol in adults with hypercholesterolaemia compared to placebo over four months.

This is a single-centre, randomised, double-blind, placebo controlled, parallel study.

Applicants will be eligible to participate if they have hypercholesterolemia, defined by fasting LDL-cholesterol 2.5mmol/L and ≤5 mmol/L confirmed at screening visit. Participants who are otherwise healthy will be included in the study; individuals with a history of cardiovascular disease are excluded from this trial.

Following pre-screening telephone assessment, applicants will attend an in-clinic screening visit and following informed consent, their general health and eligibility for inclusion into the study will be assessed.

On Day 1 eligible participants will be randomly allocated to receive one of two study treatments (intervention or placebo). Participants will consume the assigned treatment daily for four months.

Participants will return to the clinic at months 2 and 4 for assessment of primary and secondary outcomes. Compliance, adverse events and concomitant medication use will be assessed at these visits. In addition, participants will complete an online survey at months 1 and 3 to assess protocol compliance, adverse events and use of concomitant medications. Any queries that arise from the survey will be followed up by phone call.

Dietary intakes will be assessed at the baseline and four-month visits. A final participant online survey and phone call (if needed) will be conducted one month after the 4-month visit for a final safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-65 inclusive
2. Fasting LDL-cholesterol ≥2.5mmol/L and ≤5mmol/L* confirmed at screening visit
3. Low cardiovascular disease (CVD) risk score (for individuals aged 45-65 years, inclusive) determined using Framingham Risk Equation <10% absolute risk of CVD events over 5 years# as determined using a risk calculator (1) or in the event that this is not available using Australian cardiovascular risk charts (2)
4. Body mass index (BMI) >18.5 kg/m2 and <35 kg/m2 confirmed during screening period and Day 1
5. Willing to provide written Informed Consent

Exclusion Criteria:

1. Serum LDL-cholesterol >5 mmol/L* at screening
2. Use of omega-3 supplements at high dose (>900 mg/day of docosahexaenoic acid (DHA) / eicosapentaenoic acid (EPA))
3. Use of and not prepared to abstain from lipid lowering medications, supplements or fortified foods containing substances that may, in the opinion of the medical investigator, affect lipid concentrations (e.g. statins, metformin, fibrates, cholesterol absorption inhibitors, nicotinic acid, or omega-3 supplements <900 mg/day DHA/EPA) , soluble fibre, e.g. β-glucan/psyllium, plant sterols, curcumin/turmeric) within past 28 days of Day 1
4. Previous diagnosis of chronic disease such as CVD, diabetes, cancer, familial hypercholesterolaemia, kidney disease
5. Smoking (i.e. history of smoking within the last six months)
6. Serum triglycerides >4.5mmol/L (LDL-cholesterol concentrations are unreliable in the presence of high triglyceride levels)
7. Women of childbearing potential (WOCBP) who:

   1. Are not currently using effective methods of contraception and
   2. Have not been using effective methods of contraception for 14 days prior to day 1 and
   3. Are not willing to use effective methods of contraception throughout the study
8. WOCBP who have a positive urine dipstick pregnancy test at screening or Day 1, or currently pregnant or lactating
9. Untreated hypertension (blood pressure ≥140/90mmHg)
10. Aversion and/or intolerance/allergy to the study intervention products ^
11. Unwilling or unable to maintain usual levels of physical activity for the duration of the study
12. History of or known presence of alcohol abuse or illicit drug use, any surgical history, clinically significant conditions (i.e. renal, or urological disease, liver disease gastrointestinal disease or any other significant disease) or organ dysfunction that in the opinion of the investigator may affect the participant's ability to participate in the study or the study results
13. Currently hospitalised or any planned hospitalisations during the study or up to one month following the last dose of the study product that may affect the participant's ability to comply with the study in the opinion of the Medical Investigator
14. Received an investigational drug within 3 months prior to Day 1 that in the opinion of the investigator may affect the applicant's ability to participate in the study or the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Change in LDL-cholesterol | From baseline to 4 months
  Low-density lipoprotein-cholesterol (LDL-C) will be analysed using standardised methods. A Beckman AU480 clinical analyser (Beckman Coulter Inc, Brea, CA, USA) and relevant commercial enzymatic test kits will be used for analysis of serum LDL-cholesterol.
  Change in serum LDL-C (mmol/L) from baseline will be recorded.

SECONDARY OUTCOMES:
Serum lipid concentrations from baseline | From baseline to 4 months
  Change in serum lipid concentrations of the following measures (total cholesterol, high-density lipoprotein-cholesterol, triglycerides, non-HDL-C, total cholesterol:HDL-cholesterol ratio, apolipoproteinA1 (apoA1), apolipoproteinB (apoB), apoB:apoA1 ratio) will be analysed. Fasting blood samples (total of ~14 ml) will be collected into vacutainers containing a clot activator for the preparation of serum.
  Secondary blood-based outcomes will be analysed using standardised methods. Immunoturbidimetric test kits will be used for analysis of apoA1 and apoB. Total cholesterol:HDL-cholesterol and apoB:apoA1 ratio will be calculated from the results. Non-HDL-cholesterol will be calculated as total cholesterol - HDL-cholesterol.
Blood pressure changes from baseline | From baseline to 4 months
  Resting systolic and diastolic blood pressure (mmHg) will be measured using an automated blood pressure monitor in a seated position following a 5-minute rest. The average of three measurements (separated by 2 minutes) will be recorded.
Changes in HbA1c from baseline | From baseline to 4 months
  Whole Ethylenediaminetetraacetic acid (EDTA) blood samples will be collected to analyse haemoglobin A1C (HbA1c) concentration changes during the study period. A Beckman AU480 clinical analyser (Beckman Coulter Inc, Brea, CA, USA) and relevant commercial enzymatic test kits will be used for analysis of HbA1c.
Changes in plasma ox-LDL | From baseline to 4 months
  Changes in plasma oxidised-low-density lipoprotein will be analysed by commercial ELISA kit. Vacutainers containing K2-EDTA anticoagulant will be used for the preparation of plasma. This assay will be measured on an EnVision Multilabel plate reader (Perkin Elmer, MA, USA).
Changes in serum malondialdehyde | From baseline to 4 months
  Changes in serum malondialdehyde will be analysed by commercial colorimetric assay kit. This assay will be measured on an EnVision Multilabel plate reader (Perkin Elmer, MA, USA).
Changes to diet | From baseline to 4 months
  Participant's habitual dietary intake will be assessed at Baseline and 4 month visits using the Automated Self-Administered 24-hour (ASA24-Australia) Dietary Assessment Tool, version (2016), developed and validated by the National Cancer Institute, Bethesda, MD (36). Three 24-hour recalls will be completed at each occasion. At Day 1, participants will complete the first 24-hour recall during a dietitian consultation while the subsequent 24-hour recalls will be completed by the participant at home within 7-days of Day 1 and on days as specified by the dietitian (including 2 week- and 1 weekend day). Overall, all days of the week will be covered by participants. Nutrient analysis is automated through the ASA24 program and uses the Australian Food, Supplement and Nutrient Database (AUSNUT, 2011-13).
Changes in anthropometric measurements - height | From baseline to 4 months
  Height will be measured at Screening (cm). Height will be measured using a stadiometer.
  Waist and hip circumference (cm) will be measured at Baseline, 2- and 4 month or Early Withdrawal visits. Waist will be measured at the top of the iliac crest with a plastic measuring tape and taken at minimal respiration for the average of three consecutive readings. Hip circumference will be measured at the largest circumference of the buttocks.
Changes in anthropometric measurements - weight | Baseline to 4 months
  Body weight (kg) will be measured at screening and Day 1 and also be collected at the 2 month, 4 month or Early Withdrawal visits. Body weight will be measured using calibrated electronic digital scales.
Changes in anthropometric measurements - BMI | Baseline to 4 months.
  Body mass index (BMI) will be calculated using the formula weight (kg)/height (m)2. BMI will be assessed at screening, baseline, 2 months, and 4 months.
Changes in anthropometric measurements- WHR | Baseline to 4 months
  Waist:hip ratio (WHR) will be calculated using the formula waist circumference (cm)/hip circumference (cm). WHR will be calculated from measurements taken at Baseline, 2 and-4 months or Early Withdrawal visits.
Changes in body composition | From baseline to 4 months
  Fat mass and fat free mass will be measured at Baseline, 2- and 4 month or Early Withdrawal visits using a multi-frequency bioelectrical impedance analysis machine with 8 tactile electrodes (InBody 770, Biospace Co. Ltd, Seoul). Measurements will be obtained after voiding. Participants will stand upright, positioning their bare feet on the footpads and their hands on the handles. A small electrical current is passed through the body, resistance is measured, and total body water and the corresponding body composition measures are calculated by the inbuilt software.
Safety - Incidence of adverse events (AEs) and serious adverse events (SAEs) | From baseline to 4 months
  All adverse events will be recorded from dosing until the end of the study (Final Safety Visit or early withdrawal). At clinic visit at month 2 and month 4 and online surveys, participants will be questioned in a non-leading manner regarding the occurrence of any adverse medical event. All AEs will be documented in the source documents and evaluated by the Medical Investigator for severity and causality to study treatment. All SAEs will be reported to the study sponsor as per standard Good Clinical Practice (GCP) requirements.
Safety- Number of participants with significant changes to blood pressure over study period between groups | Baseline to 4 months
  Vital signs will be measured by a designee while the participant is seated. Resting blood pressure (systolic/diastolic mmHG) will be measured using an automated blood pressure monitor in a seated position following a 5-minute rest. The average of three measurements (separated by 2 minutes) will be recorded.Vital signs will be performed at Screening, Baseline, 2 month and 4 month or Early Withdrawal Visit.
Safety - Number of participants who fall pregnant (WOCBP only) | Baseline to 4 months
  A urine sample will be collected at Screening, Baseline, 2 and 4 month Visit or Early Withdrawal visit in WOCBP only. Study staff will perform a dipstick urine pregnancy test and record the result in the source documents.
Safety - Number of participants with significant changes to heart rate between groups | Baseline to 4 months
  Vital signs will be measured by a designee while the participant is seated. Heart rate will be measured as beats/minute by palpating the participants' carotid and radial pulses. Vital signs will be performed at Screening, Baseline, 2 month and 4 month or Early Withdrawal Visit.
Number of participants with changes to heart sounds | Baseline to 4 months
  The Medical Investigator will perform a non-invasive physical examination of the participants' cardiovascular system by listening to heart sounds to determine whether there is a heart murmur or irregular heart beat.
  At Day 1 (Baseline visit) these will be reviewed to establish their baseline characteristics.
  A symptom directed physical exam will be conducted at 4 months or Early Withdrawal Visit.
Safety - Number of participants with significant changes to respiratory rate between groups | Baseline to 4 months
  Respiratory rate will be measured by counting the number of times the chest rises per minute while the participant is at rest. Vital signs will be performed at Screening, Baseline, 2 month and 4 month or Early Withdrawal Visit.
Number of participants with changes to respiratory effort | Baseline to 4 months
  The Medical Investigator will perform a non-invasive physical examination of the participants' lung function by observing the participants' breathing rhythm and chest movement.
  At Day 1 (Baseline visit) these will be reviewed to establish their baseline characteristics.
  A symptom directed physical exam will be conducted at 4 months or Early Withdrawal Visit.
Safety - Number of participants with significant changes to core body temperature between groups | Baseline to 4 months
  Vital signs will be measured by a designee while the participant is seated. Body temperature (°C) will be measured using a digital thermometer.
Safety: Number of participants with macroscopic abnormalities of the eyes | Baseline to 4 months
  A non-invasive physical examination will be performed by a Medical Investigator and will include an assessment of the appearance of the pupil, iris, cornea, eyelids, eyelashes, conjuctiva and periorbital are including redness, discharge, lesions, ulcers, abrasions or unusual growths.
  At Day 1 (Baseline visit) these will be reviewed to establish their baseline characteristics.
  A symptom directed physical exam will be conducted at 4 months or Early Withdrawal Visit.
Safety -Number of participants with visual symptoms | Baseline to 4 months
  Participants will be asked to self-report on any visual symptoms or changes e.g. blurriness, eye strain etc. throughout the study period.
  At Day 1 (Baseline visit) these will be reviewed to establish their baseline characteristics.
  A symptom directed physical exam will be conducted at 4 months or Early Withdrawal Visit.
Safety: Number of participants with infections in the Ears, Nose, Mouth and Throat | Baseline to 4 months
  A non-invasive physical examination will be performed by a Medical Investigator and will include
  * A visual assessment of the ears, nose, mouth and throat to check for signs of infection
  * Palpation of the cervical chain lymph nodes to check for signs of infection
  At Day 1 (Baseline visit) these will be reviewed to establish their baseline characteristics.
  A symptom directed physical exam will be conducted at 4 months or Early Withdrawal Visit.
Safety: Number of participants with changes to peripheral vascular function | Baseline to 4 months
  A non-invasive physical examination will be performed by a Medical Investigator and will include palpating the dorsal pedis pulse, posterior tibial pulse and palpation of the ankles to check for peripheral oedema.
  At Day 1 (Baseline visit) these will be reviewed to establish their baseline characteristics.
  A symptom directed physical exam will be conducted at 4 months or Early Withdrawal Visit.
Safety: Number of participants with respiratory disease | Baseline to 4 months
  The Medical Investigator will perform a non-invasive physical examination of the participants' respiratory system by listening to breath sounds to determine whether there is untreated asthma or other lung disease.
  At Day 1 (Baseline visit) these will be reviewed to establish their baseline characteristics.
  A symptom directed physical exam will be conducted at 4 months or Early Withdrawal Visit.
Safety: Number of participants with changes to the gastrointestinal tract | Baseline to 4 months
  Medical Investigator will perform a non-invasive physical exam by observing and palpating the participants' abdomen to check for surgical scars, ascites, organomegaly and abdominal discomfort.
  At Day 1 (Baseline visit) these will be reviewed to establish their baseline characteristics.
  A symptom directed physical exam will be conducted at 4 months or Early Withdrawal Visit.
Safety: Changes to characteristics in physical examination - musculoskeletal | Baseline to 4 months
  A non-invasive physical examination will be performed by a Medical Investigator and will include an assessment of joint mobility. Participants will be asked to to stand and sit back down into a chair unassisted, to reach forward and try to touch their toes, and to touch their opposite shoulder blades across their front, behind their neck and behind their back (Apley Shoulder test).
  At Day 1 (Baseline visit) these will be reviewed to establish their baseline characteristics.
  A symptom directed physical exam will be conducted at 4 months or Early Withdrawal Visit.
Safety: Number of participants with changes to characteristics in skin appearance | Baseline to 4 months
  A non-invasive physical examination will be performed by a Medical Investigator who will observe the participants' skin colour, looking for central and peripheral cyanosis, jaundice, or any skin rashes or lesions.
  At Day 1 (Baseline visit) these will be reviewed to establish their baseline characteristics.
  A symptom directed physical exam will be conducted at 4 months or Early Withdrawal Visit.
Safety: Number of participants with clinically significant changes in biochemistry - AST | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in Aspartate aminotransferase (AST) from baseline (U/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry- ALT | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in Alanine aminotransferase (ALT) from baseline (U/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - GGT | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in gamma glutamyltransferase from baseline (U/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - ALP | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in Alkaline phosphatase (ALP) (U/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - LD | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in Lactate Dehydrogenase (U/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - creatinine | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in creatinine (µmol/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - creatinine kinase | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in creatinine kinase (U/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - urea nitrogen | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in urea nitrogen (mmol/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - sodium | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in blood sodium levels (mmol/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - potassium | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in blood potassium levels (mmol/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - chloride | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in blood chloride levels (mmol/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - bicarbonate | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in blood bicarbonate levels (mmol/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - urea | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in blood urea levels (mmol/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - calcium | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in calcium levels (mmol/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - CRP | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in C-reactive protein levels (CRP) measured as mg/L will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - uric acid | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in uric acid measured as mol/mol will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - phosphate | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in phosphate (mmol/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - albumin | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in albumin (g/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - globulins | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in globulins (g/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - protein | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in protein (g/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - total bilirubin | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in total bilirubin (umol/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in biochemistry - glucose | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in fasting glucose (mmol/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - RDW | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in red cell distribution (RDW) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - haemoglobin | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in haemoglobin (g/L) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - RBC | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in red blood cell count (RBC) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - PCV | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in packed cell volume (PCV) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - MCV | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in mean cell volume (MCV) will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - MCHC | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in mean cell hemoglobin concentrations (MCHC) measured as g/L will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - platelets | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in the number of platelets will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - white cell count (WCC) | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  Changes in the number of white cells will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - neutrophils | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  A white cell count differential test will be conducted. Changes in the number of neutrophils will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - lymphocytes | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  A white cell count differential test will be conducted. Changes in the number of lymphocytes will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - monocytes | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  A white cell count differential test will be conducted. Changes in the number of monocytes will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - eosinophils | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  A white cell count differential test will be conducted. Changes in the number of eosinophils will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.
Safety: Number of participants with clinically significant changes in haematology - basophils | Baseline to 4 months
  Fasting blood samples will be collected at Screening, Baseline, 2 Month, 4 Month and Early Withdrawal visits.
  A white cell count differential test will be conducted. Changes in the number of basophils will be analysed by a National Association of Testing Authorities, Australia (NATA) laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Welma Stonehouse, PhD, Principal Investigator — Commonwealth Scientific and Industrial Research Organisation, Australia
Locations (1):
- CSIRO Nutrition and Health Research Clinic, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stonehouse W, Benassi-Evans B, Louise J. The effects of a novel nutraceutical combination on low-density lipoprotein cholesterol and other markers of cardiometabolic health in adults with hypercholesterolaemia: A randomised double-blind placebo-controlled trial. Atherosclerosis. 2025 Apr;403:119177. doi: 10.1016/j.atherosclerosis.2025.119177. Epub 2025 Mar 22. PMID 40147213